CLINICAL TRIAL: NCT03815032
Title: Assessing the Accuracy of the OptoWire DeuxTM in a Wire to Wire Comparison
Acronym: ACCURACY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Opsens, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18.238
Record Dates: First submitted 2019-01-07; First posted 2019-01-24 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Atherosclerosis; Atherosclerosis, Coronary; Angina, Stable; Angina, Unstable; NSTEMI - Non-ST Segment Elevation MI
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Atherosclerosis; Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optowire Deux FFR assessment (1) (Experimental): A total of 45 consecutive patients will be recruited:
  group 1 (n=30): To assess the differences in FFR measurements (drift) made by the OptoWire Deux FFRTM guidewire by comparison of simultaneous data of two different OptoWire DeuxTM guidewires
  Interventions: Device: Drift assessment of OptoWire Deux FFR wire (1)
- Optowire Deux FFR assessment (2) (Experimental): group 2 (n=15): To assess the differences in FFR measurements (drift) obtained from an OptoWire DeuxTM FFR guidewire and compare it to the FFR measurement by a VERRATATM guidewire
  Interventions: Device: Drift assessment of OptoWire Deux FFR wire (2)

INTERVENTIONS:
Device: Drift assessment of OptoWire Deux FFR wire (1) — Simultaneous data of two different OptoWire DeuxTM guidewires (group 1) to assess a single coronary stenosis and detect any difference if any.
  Arms: Optowire Deux FFR assessment (1)
Device: Drift assessment of OptoWire Deux FFR wire (2) — Simultaneous data of one Optowire Deux TM guide wires and one VERRATA-TM FFR wire (group 2) to assess a single coronary stenosis and detect any difference if any.
  Arms: Optowire Deux FFR assessment (2)

SUMMARY:
The goal of the ACCURACY study is to assess the differences, if any, in FFR measurements made by the OptoWire Deux FFR guidewire by comparison of simultaneous data of two different OptoWire DeuxTM guidewires (group 1). In addition, the investigators will compare (group 2) the FFR measurements obtained from an OptoWire Deux FFR guidewire and compare it to the FFR measurement by a VERRATA-TM guidewire to assess coronary stenosis in the routine clinical practice.

DETAILED DESCRIPTION:
This is a single center, prospective, non-blinded clinical investigation enrolling consecutive patients with coronary lesion candidate for FFR assessment. The study aim to assess the differences, if any, in FFR measurements made by the OptoWire Deux FFR guidewire by comparison of simultaneous data of two different OptoWire DeuxTM guidewires (group 1, n=30). In addition, The investigators will compare (group 2, n=15) the FFR measurements obtained from an OptoWire Deux FFR guidewire and compare it to the FFR measurement by a VERRATA-TM guidewire to assess coronary stenosis in the routine clinical practice. The clinical investigation will be conducted in the Centre Hospitalier de l'Université de Montréal (CHUM). No clinical follow-up is requested after the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Single de novo coronary lesion or in-stent restenosis lesion with an operator assessed reference diameter ≥2.0 mm requiring FFR measurement based on the operator's clinical judgment

Exclusion Criteria:

* Patients with ST-segment-elevation myocardial infarction (STEMI), culprit lesion of non-ST-segment-elevation myocardial infarction (NSTEMI), New York Heart Association class IV heart failure, suspected or visible thrombus, dissection or excessive calcification or tortuosity in the target vessel, or a stenosis in a bypass graft will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
delta FFR | Day 1
  To assess the magnitude of reading delta from wire to wire in a percutaneous coronary intervention

SECONDARY OUTCOMES:
Drift recording | Day 1
  The rate of significant drift, defined as Pd/Pa <0.97 or >1.03
Delta from guidewire to guidewire | Day 1
  Assess the magnitude of reading delta from guidewire to guidewire prior to equalization.
Stents | Day 1
  The number of stents used.
Stents on FFR wire | Day 1
  The number of stents placed over an OptoWire DeuxTM guidewire.
Workhorse guidewire | Day 1
  Number of Workhorse guidewire used.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Mansour, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Pothineni NV, Shah NN, Rochlani Y, Nairooz R, Raina S, Leesar MA, Uretsky BF, Hakeem A. U.S. Trends in Inpatient Utilization of Fractional Flow Reserve and Percutaneous Coronary Intervention. J Am Coll Cardiol. 2016 Feb 16;67(6):732-733. doi: 10.1016/j.jacc.2015.11.042. No abstract available. PMID 26868697
- [Result] Fearon WF. Percutaneous coronary intervention should be guided by fractional flow reserve measurement. Circulation. 2014 May 6;129(18):1860-70. doi: 10.1161/CIRCULATIONAHA.113.004300. No abstract available. PMID 24799502